CLINICAL TRIAL: NCT04401514
Title: Does ROCKING Chairs Calm Delirious Patients in the Intensive Care Unit: a Multicenter Clinical Randomized Trial (RockingICU)
Brief Title: Does Rocking Charis Calm Delirious Patients in the Intensive Care Unit
Acronym: RocingICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scandinavian Critical Care Trials Group (Other)
Responsible Party: Principal Investigator, Anders Perner, Professor, Scandinavian Critical Care Trials Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RockingICU
Record Dates: First submitted 2019-11-04; First posted 2020-05-26 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiemntal intervention (Experimental): The experimental intervention is a 20 min. long rocking chair with music therapy.
  Interventions: Device: Rocking chair therapy
- Control intervention (Active Comparator): Control intervention is also transferred to the rocking chair, but the therapy program will not be turned on.
  Interventions: Device: Rocking chair therapy

INTERVENTIONS:
Device: Rocking chair therapy — 20 min long rocking therapy with music cure. The therapy can be extended if needed

SUMMARY:
Background: Delirium among patients admitted to an ICU is a common condition associated with increased morbidity and mortality. To this point no evidence-based prevention or treatment exist for delirium. Non-pharmacological interventions such as early mobilization and systematic bundle of care have been suggested to decrease the number of days of delirium. So far there exist no studies exploring if delirious patients benefit or not when mobilized to a rocking chair with music therapy.

Objectives: To assess if rocking chair therapy can decrease the burden of delirium in adult, critical ill patients admitted to an ICU.

Design: A clinical initiated multicenter randomized non-blinded trial, of delirious patients mobilized to a rocking chair versus no rocking chair.

Inclusion and exclusion criteria: Inclusion criteria: Adult intensive care patients (18 years and above) diagnosed with delirium with a validated screening tool. Exclusion criteria: if the patient is evaluated not to be mobilized to a rocking chair and expressing discomfort and do not wish to be mobilized, a patient with critical illness neuropati, patients with lever coma, patient in ECM treatment, patients that are mentally permanently incompetent, not receiving active life support if needed, weight more that 130 kg, if informed consent cannot be obtained, if the patient is admitted because of suicide attempt and is the patient have delirium tremens.

Intervention: The experimental intervention is a 20 min. long rocking chair with music therapy. Control intervention is also transferred to the rocking chair, but the therapy program will not be turned on. Standardized pharmacological and non-pharmacological interventions for delirium will continue for both groups. Delirium and consciousness will be evaluated twice a day.

Outcomes: Primary outcome: number of days alive without coma and delirium in the ICU. Secondary outcome: Number of days admitted to the ICU and number of patients with at least one difference in RASS score before end after the experimental intervention.

Trial size: A power calculation have estimated that a total number of 76 patients with delirium should be included in each study group.

Time schedule: We estimate that the inclusion period and follow up will as long as 1 year from the time the first patient is randomized.

Amendment's protocol Agreed by the project group August 22nd 2022, we will do an additional 90-day follow-up of all-cause mortality. This was agreed before the project group or statistician had access to the randomisation key and intervention data, and before any statistical analysis was started.

DETAILED DESCRIPTION:
The intervention is a 30 min long transfer to a rocking chair with music cure therapy. For the intervention group, the intervention will be turned on and for the control, the rocking and music function will not be turned on.

ELIGIBILITY:
Inclusion Criteria:

* admitted to ICU
* positive delirium evaluation with CAM-ICU or ICDSC

Exclusion Criteria:

* if the patient is evaluated not to be mobilized to a rocking chair
* expressing discomfort and do not wish to be mobilized
* patients with critical illness neuropathy
* patients with levercoma
* patient in ECOM (exstracorporel membrane oxygenation) treatment
* patients that are mentally permanently incompetent
* patients not receiving active life support if needed
* patients that weight more than 130 kg
* patients were informed consent cannot be obtained
* patients admitted because of suicide attempt
* patients with delirium tremens

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2022-11-13 (Actual)

PRIMARY OUTCOMES:
number of days alive without coma and delirium in the ICU | 14 day follow up

SECONDARY OUTCOMES:
Number of days admitted to the ICU | 14 day follow up
Delta RASS | 14 day follow up
  RASS score goes from +4 very agitated to -5 is coma. A score of 0 is equal to alert and calm
all cause mortality | 90 day follow up
  all cause mortality at additional follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Egerod, Professor, Study Chair — Department of Intensive care, Copenhagen University Hospital, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collet MO, Nielsen GM, Thorn L, Laerkner E, Fischer S, Bang B, Langvad A, Granholm A, Egerod I. Rocking Motion Therapy for Delirious Patients in the ICU: A Multicenter Randomized Clinical Trial. Crit Care Med. 2025 Jan 1;53(1):e161-e172. doi: 10.1097/CCM.0000000000006495. Epub 2024 Nov 15. PMID 39792532